CLINICAL TRIAL: NCT04100252
Title: The Impact of Amniotic Fluid Index (AFI) on Maternal and Perinatal Outcomes in Pregnant Women With Preterm Premature Rupture of Membranes (PPROM)
Brief Title: The Impact of Amniotic Fluid Index (AFI) on Maternal and Perinatal Outcomes in Pregnant Women With Preterm Premature Rupture of Membranes
Acronym: AFI in PPROM
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Özkan Özdamar, M.D., Associate Professor of Obstetrics and Gynecology, Istanbul Medeniyet University
Other Study IDs: 2018/0480
Record Dates: First submitted 2019-09-10; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Premature Rupture of Membrane; Amniotic Fluid Leakage; Maternal Complication of Pregnancy; Fetal Complications
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Women with AFI<5 cm at the time of PPROM diagnosis): Pregnant women who were diagnosed PPROM the gestational ages of 23+0 and 33+0 were examined ultrasonographically at the first admission. Women with AFI<5 were enrolled in the Group 1.
  Interventions: Other: AFI via transabdominal ultrasonography
- Group 2 (Women with AFI≥5 cm at the time of PPROM diagnosis): Pregnant women who were diagnosed PPROM the gestational ages of 23+0 and 33+0 were examined ultrasonographically at the first admission. Women with AFI≥5 were enrolled in the Group 2.
  Interventions: Other: AFI via transabdominal ultrasonography

INTERVENTIONS:
Other: AFI via transabdominal ultrasonography — AFI via transabdominal ultrasonography was performed at the time of diagnosis.

SUMMARY:
Pregnant women who admitted with the complaint of amniotic fluid leakage between the gestational ages of 23+0 and 33+0 and who finally were diagnosed as PPROM were included in the study. Women with multiple gestations, cervical dilatation above 6 cm at the admission, hypertensive diseases, cervical cerclage, fetal anomalies, olgohydramnios, polihydramnios, and those who declined to involve in the study were excluded.

In all included women were examined at the admission for amniotic fluid index via trans abdominal ultrasonography. AFI were measured by four quadrant technique, which is sum of the deepest vertical length of pocket of fluid in each quadrant without any umbilical cord. All included patients were assessed in two groups; women with AFI<5 and those with AFI≥5 cm.

Included patients were followed in terms of maternal and fetal complications. Maternal complications were chorioamnionitis, placental abruption, placental retention, postpartum endometritis, postpartum hemorrhage; while fetal complications comprised necessity of admission to neonatal intensive care unit, neonatal sepsis, meconium aspiration syndrome, respiratory distress syndrome, intraventricular hemorrhage, umbilical cord pH below 7.10, APGAR score of 5th minute below 5. All complication rates were compared between the groups. In addition, the time period between the diagnosis of PPROM and the time of delivery was defined as latency period and were compared between the groups.

DETAILED DESCRIPTION:
Pregnant women who admitted with the complaint of amniotic fluid leakage between the gestational ages of 23+0 and 33+0 were examined for the inclusion criteria of the study. Among them, women with usual history of gross amniotic fluid leakage as well as classical speculum findings of ROM, such as pooling of amnitotic fluid within the posterior fornix or vaginal wall, were diagnosed as PPROM and included in the study without any further investigation. In case of the absence of these findings and suspected cases, PPROM was diagnosed via placental alpha-microglobulin-1 test from the vaginal fluid. Those with positive test results were included in the study. Women with multiple gestations, cervical dilatation above 6 cm at the admission, hypertensive diseases, cervical cerclage, fetal anomalies, olgohydramnios, polihydramnios, and those who declined to involve in the study were excluded.

In all included women were examined at the admission for amniotic fluid index via trans abdominal ultrasonography. AFI were measured by four quadrant technique, which is sum of the deepest vertical length of pocket of fluid in each quadrant without any umbilical cord. All included patients were assessed in two groups; women with AFI<5 and those with AFI≥5 cm.

Included patients were followed in terms of maternal and fetal complications. Maternal complications were chorioamnionitis, placental abruption, placental retention, postpartum endometritis, postpartum hemorrhage; while fetal complications comprised necessity of admission to neonatal intensive care unit, neonatal sepsis, meconium aspiration syndrome, respiratory distress syndrome, intraventricular hemorrhage, umbilical cord pH below 7.10, APGAR score of 5th minute below 5. All complication rates were compared between the groups. In addition, the time period between the diagnosis of PPROM and the time of delivery was defined as latency period and were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women Diagnosis of PPROM between 23+0 and 33+0 gestational ages. -

Exclusion Criteria:

Multiple gestations, C Cervical dilatation above 6 cm at the admission, Hypertensive diseases, Cervical cerclage, Fetal anomalies, Oligohydramnios, Polihydramnios, Those who declined to participate in the study.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All pregnant women
Study Population: Pregnant women who were diagnosed as PPROM between 23+0 and 33+0 gestational ages.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Number of Pregnant Women experiencing Complications | Through study completion, an average of 1 year
  Adverse events emerging in included pregnant women from the time of PPROM diagnosis to the end of the postpartum 1st month
Number of fetuses and newborns experiencing complications | Through study completion, an average of 1 year
  Adverse events emerging in fetuses and neonates from the time of PPROM diagnosis to the end of the postpartum 1st month

SECONDARY OUTCOMES:
Latency Time | Through study completion, an average of 1 year
  The time period from the PPROM diagnosis to delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Goztepe Research and Training Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
To be assessed
Supporting Information: Study Protocol, CSR